CLINICAL TRIAL: NCT02649283
Title: Phase IV, Multicenter, Open Label, Non Randomized Comparative Group Study to Assess the Safety and Performance of the OrbiSymm in Subjects Referred to Contra Lateral Breast Symmetrisation Following Breast Reconstruction Post Mastectomy
Brief Title: Performance of OrbiSymm in Subjects Referred to Contra Lateral Breast Symmetrisation
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Orbix Medical Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: OX CL03
Record Dates: First submitted 2015-12-24; First posted 2016-01-07 (Estimated); Last update posted 2016-09-29 (Estimated); Status verified 2016-09

CONDITIONS: Breast Asymmetry Between Native Breast and Reconstructed Breast

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Breast symmetrisation with OrbiSymm (Other): Standard surgical intervention of up to 30 patients including placement of the OrbiSymm device
  Interventions: Device: OrbiSymm device
- Breast symmetrisation without device (Other): Standard surgical intervention of up to 30 patients without the Orbix device; only routine reduction/symmetrisation intervention
  Interventions: Procedure: Breast symmetrisation

INTERVENTIONS:
Device: OrbiSymm device — Breast symmetrisation following unilateral mastectomy and referred to contralateral symmetrisation procedure, with the OrbiSymm device, that requires reduction of at least 150grams.
  Other Names: Contralateral symmetrisation using OrbiSymm device
  Arms: Breast symmetrisation with OrbiSymm
Procedure: Breast symmetrisation — Breast symmetrisation following unilateral mastectomy and referred to contralateral symmetrisation procedure, without the OrbiSymm System, that requires reduction of at least 150grams.
  Other Names: Contralateral symmetrisation
  Arms: Breast symmetrisation without device

SUMMARY:
This is a Phase IV, multicenter, open label, non-randomized comparative group study to assess the safety and performance of the OrbiSymm system in subjects referred to contra lateral breast symmetrization involving a breast reduction following breast reconstruction post-mastectomy.

DETAILED DESCRIPTION:
The device has the CE Mark and will be used in the indication for which it is approved.

Up to 60 patients will be assigned to the study (up to 30 patients for Orbix procedure, and up to 30 patients without Orbix procedure (only routine reduction/symmetrisation). Patients will return to the clinic for follow-up at 1, 3, 6, 12 & 24 months (last visit will be optional).

ELIGIBILITY:
Inclusion Criteria:

1. Signed informed consent before any study specific tests or procedures are done.
2. Female subject between the age of 20 and 65 years old
3. Underwent breast reconstruction following unilateral mastectomy and referred to contra lateral symmetrisation procedure that requires reduction of at least 150gr (clarification: the procedure of reconstruction and symmetrisation may be performed simultaneously).
4. Breast size ≥D
5. BMI≤ 32

Exclusion Criteria:

1. Pregnant or lactating woman.
2. Subject with history of surgical procedures involving the ribs and rib cage.
3. Subject with documented osteoporosis (bone density per DEXA of less than -1.8).
4. Subject with breast implants.
5. Subject is suffering from breast carcinoma or residual malignant tumor in the side of symmetrisation.
6. Subject suffering from reconstruction failure, skin necrosis or implant infection.
7. Subject with diagnosed or suspected auto-immune disease.
8. Subject with pathologies that affect blood coagulation, immune system or any treatment interfering with them.
9. Subject with lesions due to radiation, ulceration, vascular anomalies or history of circulatory disorder.
10. Subject suffering from a progressive fibrocystic disease, considered to be pre-cancerous, without mastectomy.
11. Subject with concurrent diseases determined by the surgeon to pose unduly high risk of surgical and/or postoperative complications such as obesity, smoking, diabetes, autoimmune disease, coagulopathy, chronic lung or severe cardiovascular disease.
12. Use of drugs that might result in high surgical risk and/or significant postoperative complication, including drugs that would interfere with blood clotting.
13. Psychological instability, inappropriate attitude or motivation.
14. Subject participating or that has participated until one month prior to planned procedure, in another investigational study.

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2016-10; Primary Completion 2019-10 (Estimated); Study Completion 2019-10 (Estimated)

PRIMARY OUTCOMES:
Evaluate the long term performance OrbiSymm by measuring the stability of the symmetrisation before and after the procedure and during the follow up period. | up to 24 months
  Stability of symmetrisation as measured by comparison of patients' breast measurements before the procedure and during the FU period (measures will be taken by the surgeon in cm)

SECONDARY OUTCOMES:
Evaluate the performance OrbiSymm | up to 24 months
  Performance will be measured by comparison of patients' ptosis grade before the procedure and during the FU period (using ptosis grade scale 0-4)
Evaluate the long term safety of OrbiSymm | up to 24 months
  Demonstration of the safe implantation of the device by means of analysis of overall incidence and severity of procedure & device related adverse events after 1, 3, 6, 12 and 24 months (last visit will be optional). Summarizing the number of participants with treatment-related adverse events as assessed by CTCAE v4.0
Patient satisfaction | up to 24 months
  Patients will complete questionnaire regarding their satisfaction before the procedure and after 3, 6, 12 and 24 months (last visit will be optional).

CONTACTS AND LOCATIONS:
Overall Officials: Eyal Prof. Gur, M.D., Ph.D., Study Director — Medical Director, Orbix Medical
Locations (1):
- Instituto Nazionale dei Tumori di Roma "Regina Elena", Rome, Italy